CLINICAL TRIAL: NCT01558245
Title: Tissue Kallikrein Preventing the Restenosis After Stenting of Symptomatic MCA Atherosclerotic Stenosis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jinling Hospital, China (Other)
Responsible Party: Principal Investigator, Zhang Renliang, Clinical Professor and Associate Director of Department of Neurology, Jinling Hospital, China
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: KPRASS
Record Dates: First submitted 2011-12-14; First posted 2012-03-20 (Estimated); Last update posted 2013-09-12 (Estimated); Status verified 2013-09

CONDITIONS: Cerebrovascular Disease
Keywords: ischemic stroke; in-stent restenosis; tissue kallikrein;; the middle cerebral artery; atherosclerotic stenosis
MeSH Terms: conditions — Cerebrovascular Disorders; Ischemic Stroke | interventions — Tissue Kallikreins

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tissue kallikrein group (Experimental): Patients in this group will be prescribed with intravenous infusion of TK (0.15 PNAU/d, dissolved in 100ml saline) for 7 days after stenting and then oral administration of pancreatic kallikrein enteric-coated tablet (240U, 3/d) to the end of study. As the foundation treatment, all the enrolled patients will receive aspirin (100 mg/d), clopidogrel (75 mg/d), and atorvastatin (20 mg/d) for the first 6 months and continue with the combination of aspirin and atorvastatin at the previous dosage.
  Interventions: Drug: tissue kallikrein
- Control group (No Intervention): Patients in control group will receive foundation treatment, including aspirin (100 mg/d), clopidogrel (75 mg/d), and atorvastatin (20 mg/d) for the first 6 months and continue with the combination of aspirin and atorvastatin at the previous dosage.

INTERVENTIONS:
Drug: tissue kallikrein — Human urinary kallidinogenase can transform kininogen to bradykinin (kinin) and vasodilatory factors (kallidin)
  Other Names: Human urinary kallidinogenase (HUK)
  Arms: Tissue kallikrein group

SUMMARY:
The study aims to determine whether tissue kallikrein (TK) is efficacy for preventing the long-term in-stent restenosis (ISR) after stenting of symptomatic atherosclerotic stenosis of the middle cerebral artery (MCA) M1 segment

DETAILED DESCRIPTION:
A series of studies have confirmed the kallikrein-kinin system (KKS), including kallikrein, kininogen and kinin, plays an important role in the regulation of inflammation secondary to acute and chronic ischemic brain injury. Some researchers found that hTK gene delivery can inhibit the formation of neointimal induced by the common carotid artery ligation in mice. Further study revealed hTK gene transfection in VSMC lead to increased secretion of TK and inhibition of VSMC proliferation. In addition, it was also observed that the serum TK levels were coincident with the carotid artery stenosis. The more severe the stenosis is, the higher the serum TK level is, and the serum TK decreased after carotid artery angioplasty and stent placement. These results suggest that KKS play an important regulatory role in vascular remodeling and TK may exert a beneficial influence in the process of ISR

ELIGIBILITY:
Inclusion Criteria:

1. TIA or stroke in the MCA territory refractory to aggressive anti-platelet and regular statin therapy in 3 months
2. Symptomatic MCA M1 segment stenosis ≥ 70% confirmed with DSA
3. Successfully treated with PTAS without acute surgical complications in 12 hours after operation
4. All patients provided fully informed consent

Exclusion Criteria:

1. Using angiotensin-converting enzyme inhibitors
2. Severe cardiopulmonary dysfunction, chronic liver disease (A / G inversion, ALT increased 2-fold greater than normal), abnormal renal function (serum creatinine greater than 1.5 times normal)
3. Allergies, the history of allergy to multi-drug
4. The history of cerebral hemorrhage, brain tumors, brain trauma, cerebral embolism and other brain lesions
5. During pregnancy or breast-feeding
6. Not expected to complete follow-up

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Estimated)
Dates: Start 2011-12; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Target lesion failure | 12 months
  Patients will be evaluated at 1 month, 6 months, and 12 months after the stenting. The primary outcomes are the asymptomatic or symptomatic in-stent restenosis ≥ 50% (affirmed by digital subtraction angiography at 6 and 12 months), new stroke (ischemic and hemorrhagic) or aggravation of the previous ischemic stroke ipsilateral to the severe stenotic artery.

SECONDARY OUTCOMES:
Clinical endpoint | 12 months
  Stroke of other artery territories, myocardial infarction and vascular death will be conducted in-hospital and planned at 1 month, 6 months, and 12 months.

OTHER OUTCOMES:
Laboratory data | 12 months
  Laboratory data including bradykinin (BK), TK, platelet inhibitory rate, cGMP, cAMP, hs-CRP, TNF-α, IL-6, LDL-Ch and HDL-Ch will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Renliang Zhang, MD, Principal Investigator — Department of Neurology, Jinling Hospital, Nanjing University School of Medicine
Locations (1):
- Department of Neurology, Jinling Hospital, Nanjing University School of Medicine, Nanjing, Jiangsu, China

REFERENCES:
- [Derived] Shi R, Zhang R, Yang F, Lin M, Li M, Liu L, Yin Q, Lin H, Xiong Y, Liu W, Fan X, Dai Q, Zhou L, Lan W, Cao Q, Chen X, Xu G, Liu X. Tissue Kallikrein Prevents Restenosis After Stenting of Severe Atherosclerotic Stenosis of the Middle Cerebral Artery: A Randomized Controlled Trial. Medicine (Baltimore). 2016 Feb;95(6):e2809. doi: 10.1097/MD.0000000000002809. PMID 26871851
- [Derived] Lan W, Yang F, Liu L, Yin Q, Li M, Li Z, Sang H, Xu G, Ma M, Zhang Z, Liu Z, Liu X, Zhang R. Tissue kallikrein preventing the restenosis after stenting of symptomatic MCA atherosclerotic stenosis (KPRASS). Int J Stroke. 2014 Jun;9(4):533-5. doi: 10.1111/ijs.12229. Epub 2013 Dec 20. PMID 24354519